CLINICAL TRIAL: NCT05136742
Title: Aerobic Exercise With Diet Induces Hormonal, Metabolic, and Psychological Changes in Postmenopausal Elderly Women: a Randomized Controlled Trial
Brief Title: Aerobic Exercise With Diet Induces Hormonal, Metabolic, and Psychological Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, Cairo university faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: no: P.T.REC/012/002774
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Elderly; Hormones; Insulin Resistance; Depression
MeSH Terms: conditions — Insulin Resistance; Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise and diet program (Experimental): aerobic exercise with balanced restricted diet
  Interventions: Other: aerobic exercise and diet program
- diet program (Active Comparator): balanced restricted diet
  Interventions: Other: diet program

INTERVENTIONS:
Other: aerobic exercise and diet program — It is an interventional study in which 60 women estimated to enrol according to random allocation and assigned into two groups equal. The study group will receive aerobic exercises in addition to diet recommendations while the control group will receive diet recommendations. the aerobic exercises in form of treadmill training intensity of exercises high intensity, target heart rate (THR) will be60-70% of heart maximum (HR MAX)time of session 40 min initial 10 min warm up exercise on treadmill in low intensity and active phase20- 30 min intensity will increase until patient reach to THR then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercises 3 times per week for 12 weeks .insulin resistance will be measured by HOMA -IR index and sex hormones (estridol ,testosterone. sex hormone binding globin ) pre and post intervention and use zung self-rating depression scale to assess depression
  Arms: aerobic exercise and diet program
Other: diet program — balanced restricted diet
  Arms: diet program

SUMMARY:
PURPOSE:

to determine the effect of aerobic exercise training and diet on sex hormones , insulin resistance and depression and if is there correlation between these factors effect in postmenopausal obese women

BACKGROUND:

The practice of regular physical activity is recommended worldwide by different public health agencies for primary or secondary prevention of many health problems, including cancers. In particular, physical activity is associated with a 25 % reduction in the average risk of cardiovascular diseases among women, and this protective effect appears to be independent of menopausal status. Many interrelated biological mechanisms may underlie this association, such as the effect of physical activity on glucose metabolism, inflammation, immune function, and sex hormones. Indeed, endogenous sex hormones, particularly estrogens, seem to be involved in the initiation, promotion, and progression of tumors. Prolonged exposure to high endogenous hormone levels is considered one of the main risk factors for female breast cancer, with a relative risk of 2.00 (95 % confidence interval (CI): 1.47-2.71) for postmenopausal women with the highest estradiol levels . Several observational studies have found an inverse association between physical activity and circulating estrogen levels . This effect may be mediated by the decrease in fat mass, the main source of estrogens in postmenopausal women. It may also be mediated by the disruption of the menstrual cycle before menopause , especially when exercise is associated with low energy intakes. However, the assessment of the exposure to physical activity remains imprecise, because it is generally only possible to measure it in naturally living subjects using questionnaires

.

HYPOTHESES:

may have no Correlation between sex hormones and insulin resistance and depression in response to exercise and diet in postmenopausal obese women

RESEARCH QUESTION:

Is there Correlation between sex hormones and insulin resistance and depression in response to exercise and diet in postmenopausal obese women?

DETAILED DESCRIPTION:
It is an interventional study in which 60 women estimated to enrol according to random allocation and assigned into two groups equal. The study group will receive aerobic exercises in addition to diet recommendations while the control group will receive diet recommendations. the aerobic exercises in form of treadmill training intensity of exercises high intensity, target heart rate (THR) will be60-70% of heart maximum (HR MAX)time of session 40 min initial 10 min warm up exercises on treadmill in low intensity and active phase20- 30 min intensity will increase until patient reach to THR then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercises 3 times per week for 12 weeks .insulin resistance will be measured by HOMA -IR index and sex hormones (estridol ,testosterone. sex hormone binding globin ) pre and post intervention and use zung self-rating depression scale to assess depression

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria

* Sixty Postmenopausal women (55-65 y)
* Body mass index (BMI) ranged from 35to 39.9 kg/m2
* Postmenopausal more than 2 years

Exclusion Criteria:

* Exclusion criteria

  * women receiving weight-reduction interventions
  * taking lipid lowering drugs
  * regular medications(e.g., β-blockers, α-blockers, digoxin, diuretics, aspirin, nitrates, Presently using sex hormones)
  * having active chronic illness (e.g., rheumatoid arthritis, hyperthyroidism, and inflammatory bowel disease) and diabetes mellitus or other (unstable) endocrine-related diseases
  * cognitive impairment that will make it difficult to partake in the study
  * presence of malignant disease
  * blood donation within the last 30 days
  * Participation as a subject in any type of study or research during the prior 90 days
  * smoking

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
sex hormones | 12 weeks
  sex hormones levels by blood analysis
insulin resistance | 12 weeks
  insulin resistance by HOMA-IR
depression | 12 weeks
  depression levels by SDS scale

CONTACTS AND LOCATIONS:
Overall Officials: marwa M elsayed, Principal Investigator — cairo university faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing data with other researchers
Time Frame: 5 years after publication
Access Criteria: published journal

REFERENCES:
- [Derived] Elsayed MM, El Refaye GE, Rabiee A, Abouzeid S, Elsisi HF. Aerobic exercise with diet induces hormonal, metabolic, and psychological changes in postmenopausal obese women. Heliyon. 2022 Mar 24;8(3):e09165. doi: 10.1016/j.heliyon.2022.e09165. eCollection 2022 Mar. PMID 35368551